CLINICAL TRIAL: NCT01791322
Title: An Observational Study to Assess the Oncogenic Status of Colorectal Cancer Patients That Have Undergone Surgery
Brief Title: NovellusDx Tissue Collection Protocol
Status: Completed | Type: Observational
Sponsor: Fore Biotherapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PM 01.1
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2015-10

CONDITIONS: Patients That Have Been Diagnosed With Colorectal Cancer; Patients Eligible for Tumor Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pathology samples of tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
NovellusDx is developing a diagnostic platform for the personalized cancer therapy based on patient derived tumor tissue. The assay is able to sense activating mutations by monitoring their effect on a chip-based device.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have been diagnosed positive for colon cancer.
* available treatment follow up during cancer treatment

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have been diagnosed with cancer and are eligible for tumor biopsy will be enrolled.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Correct identification of tumor mutant genes | up to 12 month
  Correct identification of tumor mutant genes, in over 85% of the cases

CONTACTS AND LOCATIONS:
Overall Officials: Yakov Felig, Dr., Principal Investigator — Pathology lab Hadassah MC
Locations (1):
- Pathology Lab Hadassah Medical Center, Jerusalem, Israel